CLINICAL TRIAL: NCT07374003
Title: A Phase II, Single-Arm Clinical Study of Ipromlimab and Tuvonralimab Combined With Albumin-Bound Paclitaxel and Nedaplatin as Neoadjuvant Therapy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Ipromlimab and Tuvonralimab Combined With Albumin-Bound Paclitaxel and Nedaplatin as Neoadjuvant Therapy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Academician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2025-677-02
Record Dates: First submitted 2025-12-22; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced, Resectable
Keywords: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Albumin-Bound Paclitaxel; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 1. Ipromlimab and Tuvonralimab Dosage: 5 mg/kg, intravenous drip, Day 1, every 3 weeks
  2. Albumin-Bound Paclitaxel Dosage: 260 mg/m², intravenous drip, Day 1, every 3 weeks
  3. Nedaplatin Dosage: 75 mg/m², intravenous drip, Day 1, every 3 weeks
  Treatment Scheme:
  1. Neoadjuvant Therapy (2-4 cycles): Patients receive study drugs Q3W. Response is assessed after 2 cycles to decide on continuing to 4 cycles or proceeding to surgery.
  2. Surgery: Radical esophagectomy is performed within 4-6 weeks post-neoadjuvant therapy.
  3. Postoperative Management:
  pCR with R0 resection: Observation. Non-pCR with R0 resection: Adjuvant therapy. Non-R0 resection: Treatment per MDT decision.
  Interventions: Drug: lpromlimab and Tuvonralimab lpromlimab and Tuvonralimab Combined with Albumin-Bound Paclitaxel and Nedaplatin

INTERVENTIONS:
Drug: lpromlimab and Tuvonralimab lpromlimab and Tuvonralimab Combined with Albumin-Bound Paclitaxel and Nedaplatin — 1. Ipromlimab and Tuvonralimab Dosage: 5 mg/kg, intravenous drip, Day 1, every 3 weeks
  2. Albumin-Bound Paclitaxel Dosage: 260 mg/m², intravenous drip, Day 1, every 3 weeks
  3. Nedaplatin Dosage: 75 mg/m², intravenous drip, Day 1, every 3 weeks
  Treatment Scheme:
  1. Neoadjuvant Therapy (2-4 cycles): Patients receive study drugs Q3W. Response is assessed after 2 cycles to decide on continuing to 4 cycles or proceeding to surgery.
  2. Surgery: Radical esophagectomy is performed within 4-6 weeks post-neoadjuvant therapy.
  3. Postoperative Management:
  pCR with R0 resection: Observation. Non-pCR with R0 resection: Adjuvant therapy. Non-R0 resection: Treatment per MDT decision

SUMMARY:
This is a Phase II, single-arm clinical study designed to evaluate the efficacy and safety of Ipromlimab combined with Tuvonralimab, plus Albumin-Bound Paclitaxel and Nedaplatin, as neoadjuvant therapy for patients with locally advanced resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Eligible patients will receive 2-4 cycles of the combined neoadjuvant therapy (administered every 3 weeks), with response assessed after 2 cycles to determine whether to continue to 4 cycles or proceed to radical esophagectomy. Postoperative management will be tailored based on pathological results: observation for patients achieving pathological complete response (pCR) with R0 resection, adjuvant therapy for non-pCR with R0 resection, and treatment per multidisciplinary team (MDT) decision for non-R0 resection. The primary objective is to assess the pathological complete response (pCR) rate, and secondary objectives include evaluating objective response rate (ORR), disease control rate (DCR), major pathological response (MPR) rate, event-free survival (EFS), disease-free survival (DFS), 3-year disease-free survival rate, overall survival (OS), and safety profile. Exploratory objectives involve identifying predictive biomarkers for neoadjuvant immunotherapy response through multi-omics analysis of biological samples. This study aims to provide evidence for optimizing neoadjuvant treatment strategies in locally advanced resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* No prior treatment for the condition.
* Diagnosis of squamous cell carcinoma confirmed by endoscopic biopsy, with agreement to provide a pre-treatment tissue sample.
* Patients must have thoracic esophageal cancer only. The primary site is determined by the center of the mass:

  1. Upper thoracic esophagus: From the thoracic inlet to the lower border of the aortic arch, corresponding to 20-25 cm from the incisors by endoscopy.
  2. Middle thoracic esophagus: From the lower border of the aortic arch to the level of the inferior pulmonary veins, corresponding to 25-30 cm from the incisors by endoscopy.
  3. Lower thoracic esophagus: From the level of the inferior pulmonary veins to the stomach, including the gastroesophageal junction, corresponding to 30-40 cm from the incisors by endoscopy.
* Deemed to have potentially resectable disease, with clinical stage III (cT3N1M0 to cT1-3N2M0) according to the UICC/AJCC TNM Staging System, 8th Edition.
* Age ≥18 years and ≤75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, meeting the following criteria (without transfusion or hematopoietic growth factor support within 14 days prior to the first dose):

  1. Hematology: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; Platelet count ≥100 × 10⁹/L; Hemoglobin ≥9.0 g/dL.
  2. Biochemistry: Total bilirubin <1.5 × upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 × ULN; Serum creatinine ≤1.5 × ULN or calculated creatinine clearance ≥50 mL/min.
  3. Coagulation: International normalized ratio (INR) ≤1.5; Activated partial thromboplastin time (APTT) ≤1.5 × ULN.
* Male and female participants of childbearing potential must agree to use medically approved contraceptive methods during the study period and for 6 months after the last dose of the study drug(s).
* The subject is capable of understanding, able to comply with study and follow-up procedures, and voluntarily signs a written informed consent form.

Exclusion Criteria:

* Disease assessed as unresectable based on imaging such as contrast-enhanced CT of the chest/abdomen, neck lymph node ultrasound, whole-body PET-CT scan (optional), or endobronchial ultrasound (EBUS) (optional). This includes: the presence of bulky lymph nodes (≥7 suspicious lymph nodes), multi-station lymph node involvement (≥2 stations of suspicious lymph nodes), or distant metastasis.
* History of other malignancies (except for cervical carcinoma in situ or cured, localized basal cell carcinoma of the skin).
* History of autoimmune diseases.
* Recent or current use of corticosteroids or immunosuppressants.
* History of severe hypersensitivity to antibody-based drugs.
* History of chronic or recurrent autoimmune diseases.
* History of interstitial lung disease, pulmonary fibrosis, diverticulitis, or systemic ulcerative gastritis.
* Documented history of congestive heart failure, angina pectoris poorly controlled by medication; ECG-confirmed transmural myocardial infarction; uncontrolled hypertension; clinically significant valvular disease; high-risk or uncontrolled arrhythmias.
* Severe systemic concurrent diseases, such as active infection or poorly controlled diabetic complications; coagulation disorders; bleeding tendency; or insufficient thrombolytic/anticoagulant therapy.
* Female participants with a positive serum pregnancy test or who are breastfeeding, or individuals of childbearing potential unwilling to use contraception during the study period.
* Active infection with HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), or positive HIV serology; or positive HBV DNA/HCV RNA.
* Allergy to any of the drugs used in this study.
* History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation).
* History of peripheral nervous system disease, significant psychiatric disorder, or central nervous system disease.
* Concurrent use of other anti-tumor drugs.
* Current participation in, or prior participation in, another clinical trial that could potentially impact the results of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
PCR | Pathologic Complete Response(pCR) Rate Defined as the proportion of participants with no residual viable tumor cells in the resected surgical specimen. ITime Frame: assessed up to 30 days post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sub-i, Guangdong, GUANGZHOU, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (lCF)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data can be shared when the study is finished and ready for publication.
Access Criteria: PI
URL: http://None

REFERENCES:
- See also: China Clinical Research Registration — https://www.medicalresearch.org.cn/cas/sso/login?clientId=9001&redirectUri=https%3A%2F%2Fwww.medicalresearch.org.cn%2Flogin
- Available data/document: Study Protocol — https://www.medicalresearch.org.cn/cas/sso/login?clientId=9001&redirectUri=https%3A%2F%2Fwww.medicalresearch.org.cn%2Flogin — China Clinical Research Registration